CLINICAL TRIAL: NCT02268890
Title: Pharmacokinetic Study of Bortezomib (VELCADE) Administered Intravenously in Taiwanese Patients With Multiple Myeloma - A Post Approval Commitment Study
Brief Title: A Pharmacokinetic Study of Bortezomib in Taiwanese Participants With Multiple Myeloma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR104583; 26866138MMY4073 (Other: Johnson & Johnson Taiwan Ltd.)
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bortezomib; Velcade
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib (Experimental): Participants will receive a 1.3 milligram per square meter per dose (mg/m^2/dose) of bortezomib intravenously on Days 1, 4, 8, and 11.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Participants will receive a 1.3 milligram per square meter per dose (mg/m^2/dose) of bortezomib intravenously on Days 1, 4, 8, and 11.
  Other Names: Velcade

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (PK-the study of the way a drug enters and leaves the blood and tissues over time) characteristics of bortezomib when administered intravenously in Taiwanese participants with multiple myeloma (cancer of the types of cells normally found in bone marrow).

DETAILED DESCRIPTION:
This is a Phase 4, single-arm, open-label (all knew the intervention of study), and multicenter (when more than 1 hospital or medical school team work on a medical research study) study to explore the pharmacokinetics with relapsed (the return of a medical problem) or refractory (not responding to treatment) multiple myeloma. The study consists of a Screening phase and a bortezomib treatment phase with defined PK sample collection time points. Participants will receive bortezomib intravenous injection two times a week up to 2 weeks (on Days 1, 4, 8, and 11) and followed by a 10-day resting phase (Days 12 to 21) for 1 treatment cycle. Pharmacokinetics will primarily be evaluated. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma based on the standard criteria
* Measurable, secretory multiple myeloma is defined as serum monoclonal immunoglobulin (Ig) G of >= 10 gram per liters (g/L), serum monoclonal IgA or IgE greater than or equal to (>=) 5 g/L, serum monoclonal IgD >= 0.5 g/L, or serum monoclonal IgM present (regardless of level), or urine M protein of >= 200 mg/24 hour at any time point of prior treatment
* Relapse or progression of myeloma following prior systemic antineoplastic therapy and meet the indication which had been approved in the drug leaflet. Relapse is defined as: a) reappearance of measurable disease (as defined above) following complete response (CR); b) >= 25 percent (%) increase in serum or urine M-protein according to IMWG (International Myeloma Working group) criteria; c) development of new or worsening lytic bone disease; d) new plasmacytomas or >=50% increase in the longest dimension of an existing plasmacytoma; e) worsening hypercalcemia (corrected serum calcium >11.5 milligram per deciliters [mg/dL-2.8 millimoles per liters [mmol/L] due to multiple myeloma
* Karnofsky performance status >=70%
* Platelet count >=50 × 10^9 /L without transfusion support within 7 days before the laboratory test

Exclusion Criteria:

* More than 3 previous lines of therapy (separate lines of therapy are defined as single or combination therapies that are either separated by disease progression or by a >6 month treatment-free interval)
* Peripheral neuropathy or neuropathic pain of National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 Grade >=2
* Any of the following within 3 weeks prior to enrollment in the study: antineoplastic or experimental therapy, corticosteroid use above 10 mg/day (prednisone or equivalent), or plasmapheresis
* Any of the following within 2 weeks prior to enrollment in the study: radiation therapy, major surgery (kyphoplasty is not considered major surgery)
* Prior malignancy other than multiple myeloma diagnosed or treated within the last 2 years, with the exception of completely resected carcinoma in situ or basal/squamous carcinoma of the skin

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Initial Observed Plasma Drug Concentration (Co) | 72 hours pre-dose on Day 1 (Baseline); post-dose on Day 11, 12, 13 and 14
  Initial concentration extrapolated to time zero (Co) will be evaluated.
Maximum Observed Plasma Concentration (Cmax) | 72 hours pre-dose on Day 1 (Baseline); post-dose on Day 11, 12, 13 and 14
  Maximum observed plasma concentration (Cmax) will be observed.
Area Under Plasma Concentration-Time Curve From Time 0 to Last Quantifiable Time Point | 72 hours pre-dose on Day 1 (Baseline); post-dose on Day 11, 12, 13 and 14
  Area under the plasma concentration-time curve from time 0 to the time of last quantifiable time point, calculated by linear trapezoidal summation.
Area Under Plasma Concentration-Time Curve From Time 0 to Infinity (AUC-Infinity) | 72 hours pre-dose on Day 1 (Baseline); post-dose on Day 11, 12, 13 and 14
  Area under the plasma concentration-time curve from time 0 to infinity, calculated as AUClast + Clast/lamda(z), where Clast is the last measurable plasma concentration and lamda(z) is the terminal rate constant.
Terminal Half-life (t1/2) | 72 hours pre-dose on Day 1 (Baseline); post-dose on Day 11, 12, 13 and 14
  Terminal half-life, calculated by 0.693/lamda(z).
Terminal rate constant (lamda[z]) | 72 hours pre-dose on Day 1 (Baseline); post-dose on Day 11, 12, 13 and 14
  Terminal rate constant estimated by log-linear regression analysis of the terminal phase of the plasma concentration versus time curve for at least 3 points.
Systemic clearance (CL) | 72 hours pre-dose on Day 1 (Baseline); post-dose on Day 11, 12, 13 and 14
  Systemic clearance after IV dose, estimated by dividing the total administered dose by the plasma (AUC-Infinity).
Apparent Volume of Distribution (Vd) | 72 hours pre-dose on Day 1 (Baseline); post-dose on Day 11, 12, 13 and 14
  Apparent volume of distribution (Vd) based on the terminal phase after intravenous administration, calculated as Dose/(Lamda[z] * AUC-Infinity).

CONTACTS AND LOCATIONS:
Locations (6):
- Taiwan (6):
  - Changhua
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District

REFERENCES:
- See also: Pharmacokinetic Study of Bortezomib (VELCADE®) Administered Intravenously in Taiwanese Patients with Multiple Myeloma - A Post Approval Commitment Study — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=7393&filename=CR104583_CSR.pdf